CLINICAL TRIAL: NCT04216004
Title: Dairy Food Consumption and Its Effects on Inflammation and the Postprandial Regulation of Muscle Protein Synthesis
Brief Title: Anti-Inflammatory Milk Matrix
Acronym: AIMM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nicholas Burd, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20173
Record Dates: First submitted 2019-12-05; First posted 2020-01-02 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Skeletal Muscle; Inflammation
MeSH Terms: conditions — Obesity; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full-fat dairy (Experimental): 3x daily servings (cup-eq) of full-fat (3.25%) commercial cow's milk.
  Interventions: Behavioral: Controlled-Feeding Intervention; Other: Full-fat milk
- Non-fat diary (Active Comparator): 3x daily servings (cup-eq) of non-fat (0%) commercial cow's milk.
  Interventions: Behavioral: Controlled-Feeding Intervention; Other: Fat-free milk
- Non-dairy control (Placebo Comparator): 3x daily servings (cup-eq) of non-dairy sourced macronutrient composition of full-fat milk.
  Interventions: Behavioral: Controlled-Feeding Intervention; Dietary Supplement: Non-dairy beverage

INTERVENTIONS:
Behavioral: Controlled-Feeding Intervention — All energy-containing food and beverages will be provided for 1-week as a controlled-feeding study.
Dietary Supplement: Non-dairy beverage — Isolated amino acid, fatty acid, and monosaccharide beverage matched to the macronutrient content of 8 fl oz whole milk.
  Arms: Non-dairy control
Other: Full-fat milk — 3 daily servings (cup-eq) of full-fat (3.25%) commercial cow's milk.
  Arms: Full-fat dairy
Other: Fat-free milk — 3 daily servings (cup-eq) of fat-free (0%) commercial cow's milk.
  Arms: Non-fat diary

SUMMARY:
Obesity is pro-inflammatory, impairs metabolism, and physically limiting. Specifically, muscle in obese persons does not synthesize proteins normally. This further increases metabolic and physical dysfunction. As such, obesity programs should not only focus on weight loss, but muscle metabolic health. Dairy nutrients have anti-inflammatory and anabolic properties, but mostly evaluated in isolation and/or pre-clinical designs. Also, it is unknown if the circulating benefits extend to the muscle. We hypothesize that dairy full-fat milk will improve these obesity characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI, body mass index ≥30, <40 kg•m-2)
* Age 40-59
* Pre-menopausal
* Sedentary/insufficiently active for prior 6 months (mo)
* Weight stable for prior 6 mo

Exclusion Criteria:

* Tobacco, nicotine (patch/gum) use (previous 6 mo)
* Alcohol consumption >10 drinks per week
* Metabolic disorders (e.g., Metabolic Syndrome, Diabetes, thyroid diseases)
* Cardiovascular disease, arrhythmias
* Hypogonadism
* Asthma
* History of uncontrolled hypertension
* Orthopedic injury/surgery (within 1 yr)
* Hepatorenal, musculoskeletal, autoimmune, or neurological disease
* History of neuromuscular problems
* Previous participation in amino acid tracer studies
* Predisposition to hypertrophic scarring or keloid formation
* Consumption of ergogenic-levels of dietary supplements that may affect muscle mass (e.g., creatine, HMB), insulin-like substances, or anabolic/catabolic pro-hormones (e.g., DHEA) within 6 weeks prior to participation
* Consumption of thyroid, androgenic, or other medications known to affect endocrine function
* Consumption of medications known to affect protein metabolism (e.g., prescription-strength corticosteroids, non-steroidal anti-inflammatories, or acne medication)
* Pregnancy
* Allergy to dairy product or lactose intolerance
* Fasting plasma glucose (FPG) ≥ 126 mg/dL
* Oral glucose tolerance test (OGTT) ≥ 200 mg/dL

Ages: 40 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Fractional synthetic rate of myofibrillar proteins by stable isotope infusion. | 0-5 hours postprandial observation period to ingesting 2 servings of respective Arm.
  Refers to rate of building new proteins in skeletal muscle contractile protein fraction. Myofibrillar protein synthesis rates will be assessed during stable isotope infusion whereby participants will ingest 2 servings of their respective dairy treatment and the postprandial response is compared between the Arms.
Blood inflammation markers by flow cytometry. | 1 week observation period to respective Arm within a controlled-feeding intervention.
  Measurement of blood cytokines, monocytes, and macrophages by flow cytometry before and after 1-week of 3 daily servings of respective dairy treatment within a controlled-feeding intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Freer Hall, Urbana, Illinois, United States